CLINICAL TRIAL: NCT01666509
Title: A Post Marketing Clinical Follow-up, Randomised, Double-blind Study Comparing the Efficacy and Tolerability of Topical Rossoseq™ With Vehicle in Rosacea Subtype 1 (Erythematotelangiectatic)
Brief Title: Efficacy and Tolerability of Topical Rossoseq™ Compared to Vehicle in Rosacea Subtype 1 (Erythematotelangiectatic)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PBB Entrepreneur Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL-068-IV-01
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Rosacea Subtype 1 (Erythematotelangiectatic)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rossoseq™ (Experimental): Gel, topically applied twice daily
  Interventions: Device: Rossoseq™
- Vehicle (Placebo Comparator): Gel, topically applied twice
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Rossoseq™
  Arms: Rossoseq™
Device: Placebo
  Arms: Vehicle

SUMMARY:
Rossoseq™ is registered for the treatment of inflammatory skin conditions. Rosacea is one such inflammatory skin disorder that has not been studied yet for the use of Rossoseq™. Whilst rosacea is showing features of an inflammatory skin disorder [1], particularly stage 1 is poorly understood and treatment options are limited and therefore this study - within the target indication - will contribute to the learning about rosacea.

DETAILED DESCRIPTION:
Male or female subjects ≥18 and < 85 years with a clinically diagnosed rosacea subtype 1 (erythematotelangiectatic) defined by a score of 6-15 for the primary and secondary features of the rosacea standard grading system (RSGS; Wilkin et al, 2004) will be enrolled.

The study will consist of a Screening visit, Baseline visit (Week 0), a telephone call at Week 1, visits at Week 2 and 4, and a follow-up telephone call at Week 5. Eligible subjects may or may not be using medication for their rosacea at the time of screening. Subjects with concomitant use of rosacea treatments will be taken off their current medication and will return for a Baseline Visit at the end of the wash-out period.

Eligible subjects will be stratified by gender at a ratio of 4:1 (Female: Male). Within the strata, subjects will be randomised at Baseline in a 2:1 ratio in favour of Rossoseq™ to receive either Rossoseq™ or vehicle.

Efficacy will be evaluated using subject rating of the rosacea specific quality of life instrument (R-QOL; Nicholson et al, 2007) during office visits and applied over the phone during the week 1 and follow-up telephone call at Week 5. An investigator rating will be performed using a "0=absent" to "3=severe" grading of the RSGS primary features flushing, nontransient erythema, papules and pustules, telangiectasia and the secondary features burning or stinging, plaques, dry appearance, edema, ocular manifestations and phymatous changes during the office visits. Ocular manifestations and phymatous changes need to be absent to be eligible for the study.

Photographs to document treatment effects will be taken at screening, baseline, week 2 and week 4.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent prior to any study-mandated procedure
* Clinically diagnosed rosacea defined by a score of ≥6 and ≤15 out of a maximum score of 30 for the primary and secondary features of the RSGS
* Female subjects of childbearing potential must be using appropriate birth control

Main exclusion Criteria:

* Pregnancy or lactation
* Women with the following menopausal symptoms within the last two years prior to screening: excessive sweating, flushing, mood changes
* Ocular manifestations of rosacea
* Peripheral location(s) of rosacea
* Phymatous changes
* Severe facial skin dryness or xerosis
* Keratoconjunctivitis sicca
* Flushing due to conditions other than rosacea
* Any other abnormal facial skin conditions, e.g., eczema, perioral dermatitis, broken and bleeding skin on area of application
* Malignancy within the past 2 years with the exception of in situ removal of basal cell carcinoma

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Symptom construct of the R-QOL | Change from baseline to Week 4
  The symptom construct contains 7 symptom related items scored by the subject as ''never'', ''rarely'', ''sometimes'', ''often'' or ''all the time''. The responses are recorded on a 1 (never)-to-5 (all the time) scale. A subject's score is the average of his or her responses to the items in the construct (1-5).

SECONDARY OUTCOMES:
Total R-QOL | Change from baseline to Week 4
  The total R-QOL is the average of all responses
Function construct of the R-QOL | Change from baseline to Week 4
Emotion construct of the R-QOL | Change from baseline to Week 4
Total RSGS score | Change from baseline to Week 4

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Study site 5, Bochum
  - Study site 2, Dülmen
  - Study Site 1, Münster
  - Study site 4, Paderborn